CLINICAL TRIAL: NCT03257904
Title: International Prospective Observational StudY on iNtrAcranial PreSsurE in Intensive Care (ICU) (SynapseICU)
Brief Title: iNtrAcranial PreSsurE in Intensive Care (ICU) (SynapseICU)
Acronym: SynapseICU
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Giuseppe Citerio, MD, Professor, University of Milano Bicocca
Other Study IDs: SynapseICU
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage; Intracerebral Hemorrhage
Keywords: intracranial pressure
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: intracranial pressure monitoring — measurement of intracranial pressure

SUMMARY:
Intracranial pressure (ICP) monitoring is the most common neuromonitoring modality used in neurocritical care units (NCCU) around the world. Uncertainties remain around intracranial pressure monitoring both in traumatic and non-traumatic brain injury, and variation in clinical practice of intracranial pressure monitoring exists between neurocritical care units.

The objectives of the study will explore intracranial pressure monitoring variation in practice to prioritise uncertainties in the clinical management of critical care patients with acute brain injury and support further collaborative hypotheses-based prospective studies.

DETAILED DESCRIPTION:
Intracranial pressure (ICP) monitoring is the most common neuromonitoring modality used in neurocritical care units (NCCU) around the world. Uncertainties remain around intracranial pressure monitoring both in traumatic and non-traumatic brain injury, and variation in clinical practice of intracranial pressure monitoring exists between neurocritical care units.

The objectives of the study will explore intracranial pressure monitoring variation in practice to prioritise uncertainties in the clinical management of critical care patients with acute brain injury and support further collaborative hypotheses-based prospective studies.

Sample Size: This international prospective observational study aims to recruit >2000 patients in coma after acute traumatic and non-traumatic brain damage admitted to >200 Intensive Care Units.

Inclusion Criteria:

* Acute brain injury (ABI) admitted to ICU following:

  1. Hemorrhagic stroke, including intracerebral hematoma and subarachnoid hemorrhage,
  2. Traumatic brain injury (penetrating and non-penetrating).
* Age >18 years old
* Glasgow Coma Score with Eyes response = 1 (no eyes opening) and Motor score ≤5 (not following commands) at the admission to ICU or neuro-worsening within the first 48 hours with no eye opening and the Motor score decreased to ≤5

Exclusion Criteria:

* ABI who are not admitted to ICU;
* ABI due to infections of the central nervous system, ischemic stroke or other causes not defined in the inclusion criteria

Outcome measures:

Glasgow Outcome Score-Extended at 6 months

Endpoint:

The primary endpoint is the variation in clinical practice around ICP monitoring in acute brain injury patients.

Screening and recruitment: 12 weeks at each centre, or the duration required to enrol 90 patients per centre.

Follow-up: outcome measures will be collected at 6 months.

Duration of study: 2 years.

The SYNAPSE-ICU study is partly funded by ESICM (ESICM Trials Group Portfolio).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Diagnosis of an acute brain injury (ABI) due to primary hemorrhagic stroke (including intracranial hemorrhage or subarachnoid hemorrhage) or traumatic brain injury;
3. Glasgow Coma Score with Eyes response = 1 (no eyes opening) and Motor score ≤5 (not following commands) at the admission to ICU or neuro-worsening within the first 48 hours with no eye opening and the Motor score decreased to ≤5.

Exclusion Criteria:

1. Acute Brain Injury (ABI) who are not admitted to ICU;
2. ABI due to infections of the central nervous system, ischaemic stroke or other causes not defined in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemorrhagic stroke, including intracerebral hematoma and subarachnoid hemorrhage, Traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 2395 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Long-term outcome measures of neurological disability | 6 months
  Extended Glasgow Outcome Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, Principal Investigator — University Milano Bicocca
Locations (1):
- ASST-Monza, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stocchetti N, Carbonara M, Citerio G, Ercole A, Skrifvars MB, Smielewski P, Zoerle T, Menon DK. Severe traumatic brain injury: targeted management in the intensive care unit. Lancet Neurol. 2017 Jun;16(6):452-464. doi: 10.1016/S1474-4422(17)30118-7. PMID 28504109
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Cnossen MC, Scholten AC, Lingsma HF, Synnot A, Tavender E, Gantner D, Lecky F, Steyerberg EW, Polinder S. Adherence to Guidelines in Adult Patients with Traumatic Brain Injury: A Living Systematic Review. J Neurotrauma. 2021 Apr 15;38(8):1072-1085. doi: 10.1089/neu.2015.4121. Epub 2016 Aug 25. PMID 26431625
- [Background] Helbok R, Olson DM, Le Roux PD, Vespa P; Participants in the International Multidisciplinary Consensus Conference on Multimodality Monitoring. Intracranial pressure and cerebral perfusion pressure monitoring in non-TBI patients: special considerations. Neurocrit Care. 2014 Dec;21 Suppl 2:S85-94. doi: 10.1007/s12028-014-0040-6. PMID 25208677
- [Background] Chesnut RM, Bleck TP, Citerio G, Classen J, Cooper DJ, Coplin WM, Diringer MN, Grande PO, Hemphill JC 3rd, Hutchinson PJ, Le Roux P, Mayer SA, Menon DK, Myburgh JA, Okonkwo DO, Robertson CS, Sahuquillo J, Stocchetti N, Sung G, Temkin N, Vespa PM, Videtta W, Yonas H. A Consensus-Based Interpretation of the Benchmark Evidence from South American Trials: Treatment of Intracranial Pressure Trial. J Neurotrauma. 2015 Nov 15;32(22):1722-4. doi: 10.1089/neu.2015.3976. Epub 2015 Aug 31. PMID 26061135
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Chesnut R, Videtta W, Vespa P, Le Roux P; Participants in the International Multidisciplinary Consensus Conference on Multimodality Monitoring. Intracranial pressure monitoring: fundamental considerations and rationale for monitoring. Neurocrit Care. 2014 Dec;21 Suppl 2:S64-84. doi: 10.1007/s12028-014-0048-y. PMID 25208680
- [Background] Le Roux P, Menon DK, Citerio G, Vespa P, Bader MK, Brophy GM, Diringer MN, Stocchetti N, Videtta W, Armonda R, Badjatia N, Boesel J, Chesnut R, Chou S, Claassen J, Czosnyka M, De Georgia M, Figaji A, Fugate J, Helbok R, Horowitz D, Hutchinson P, Kumar M, McNett M, Miller C, Naidech A, Oddo M, Olson D, O'Phelan K, Provencio JJ, Puppo C, Riker R, Robertson C, Schmidt M, Taccone F; Neurocritical Care Society; European Society of Intensive Care Medicine. Consensus summary statement of the International Multidisciplinary Consensus Conference on Multimodality Monitoring in Neurocritical Care : a statement for healthcare professionals from the Neurocritical Care Society and the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Sep;40(9):1189-209. doi: 10.1007/s00134-014-3369-6. Epub 2014 Aug 20. PMID 25138226
- [Background] Stocchetti N, Maas AI. Traumatic intracranial hypertension. N Engl J Med. 2014 Sep 4;371(10):972. doi: 10.1056/NEJMc1407775. No abstract available. PMID 25184881
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Background] Cossu G, Messerer M, Stocchetti N, Levivier M, Daniel RT, Oddo M. Intracranial pressure and outcome in critically ill patients with aneurysmal subarachnoid hemorrhage: a systematic review. Minerva Anestesiol. 2016 Jun;82(6):684-96. Epub 2016 Apr 5. PMID 27045637
- [Background] Citerio G, Oddo M, Taccone FS. Recommendations for the use of multimodal monitoring in the neurointensive care unit. Curr Opin Crit Care. 2015 Apr;21(2):113-9. doi: 10.1097/MCC.0000000000000179. PMID 25689123
- [Background] Stocchetti N, Le Roux P, Vespa P, Oddo M, Citerio G, Andrews PJ, Stevens RD, Sharshar T, Taccone FS, Vincent JL. Clinical review: neuromonitoring - an update. Crit Care. 2013 Jan 15;17(1):201. doi: 10.1186/cc11513. PMID 23320763
- [Derived] Robba C, Graziano F, Guglielmi A, Rebora P, Galimberti S, Taccone FS, Citerio G; SYNAPSE-ICU Investigators. Treatments for intracranial hypertension in acute brain-injured patients: grading, timing, and association with outcome. Data from the SYNAPSE-ICU study. Intensive Care Med. 2023 Jan;49(1):50-61. doi: 10.1007/s00134-022-06937-1. Epub 2023 Jan 9. PMID 36622462
- [Derived] Dallagiacoma S, Robba C, Graziano F, Rebora P, Hemphill JC, Galimberti S, Citerio G; SYNAPSE-ICU Investigators. Intracranial Pressure Monitoring in Patients With Spontaneous Intracerebral Hemorrhage: Insights From the SYNAPSE-ICU Study. Neurology. 2022 Jul 12;99(2):e98-e108. doi: 10.1212/WNL.0000000000200568. Epub 2022 May 4. PMID 35508390
- [Derived] Robba C, Graziano F, Rebora P, Elli F, Giussani C, Oddo M, Meyfroidt G, Helbok R, Taccone FS, Prisco L, Vincent JL, Suarez JI, Stocchetti N, Citerio G; SYNAPSE-ICU Investigators. Intracranial pressure monitoring in patients with acute brain injury in the intensive care unit (SYNAPSE-ICU): an international, prospective observational cohort study. Lancet Neurol. 2021 Jul;20(7):548-558. doi: 10.1016/S1474-4422(21)00138-1. PMID 34146513
- [Derived] Citerio G, Prisco L, Oddo M, Meyfroidt G, Helbok R, Stocchetti N, Taccone F, Vincent JL, Robba C, Elli F, Sala E, Vargiolu A, Lingsma H. International prospective observational study on intracranial pressure in intensive care (ICU): the SYNAPSE-ICU study protocol. BMJ Open. 2019 Apr 20;9(4):e026552. doi: 10.1136/bmjopen-2018-026552. PMID 31005932